CLINICAL TRIAL: NCT01801137
Title: A Multicentre Phase III Trial to Determine the Efficacy of RAD 001 (Everolimus, Afinitor) as Second Line Therapy in Patients With Transitional Cell Carcinoma TCC of the Urothelium Which Failed or Progressed After First Line Chemotherapy
Brief Title: The Efficacy of RAD 001 as Second Line Therapy in Patients With Transitional Cell Carcinoma TCC of the Urothelium
Acronym: AFINIVEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/23
Record Dates: First submitted 2013-02-12; First posted 2013-02-28 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — Everolimus

ARMS (1):
- Afinitor (Experimental): Treatment by Afinitor 10 mg per day
  Interventions: Drug: Everolimus (Afinitor®)

INTERVENTIONS:
Drug: Everolimus (Afinitor®)

SUMMARY:
A study to determine the efficacy of Everolimus(Afinitor®) as third line therapy in patients with transitional cell carcinoma of the urothelium which failed or progressed after two lines of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male or female aged more than 18 years
* Histologically proven transitional cell carcinoma of the urothelium
* Metastatic or locally advanced disease not amenable to curative surgery and/or radiotherapy
* Recurrence or progression after at least one chemotherapy regimen and for unresectable/advanced disease
* No more than 2 lines of previous chemotherapy..
* Measurable disease (RECIST criteria)
* Previously irradiated lesions are not considered measurable- ECOG performance status of 0, 1 or 2

Exclusion Criteria:

* No prior treatment with anti cancer agents, including radiotherapy, in the last 4 weeks.
* No currently active CNS involvement
* No pregnancy. Women of child bearing potential must have a negative pregnancy test.
* No uncontrolled diabetes
* No symptomatic coronary artery disease, myocardial infarction within the last six months, congestive cardiac failure greater than New York Heart Association (NYHA) class II, uncontrolled or symptomatic cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 12 weeks | 3 months
  If a patient has not had an event, Progression-free survival is censored at the date of last adequate tumor assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital FOCH, Suresnes, Île-de-France Region, France